CLINICAL TRIAL: NCT03865667
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Preserve Femoral Stem
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002G
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Total Hip Arthroplasty: Single-arm, single-center, prospective follow-up study with consecutively enrolled newly or previously implanted subjects with the PROFEMUR® Preserve Femoral Stem(s) and CoCr (cobalt-chromium) Modular Neck combined with other Wright Medical Technologies (WMT) or MPO (MicroPort) THA (Total Hip Arthroplasty) components including acetabular shells, acetabular liners and femoral heads.
  Interventions: Device: PROFEMUR® Preserve Femoral Stem

INTERVENTIONS:
Device: PROFEMUR® Preserve Femoral Stem — Total Hip Total Hip Arthroscopy

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in Europe. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Newly or previously implanted subjects must meet all the following inclusion Criteria:

* Has undergone primary Total Hip Arthroscopy for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;lnflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity;
* Subject is implanted with the PROFEMUR® Preserve Femoral Stem(s) and cobalt-chromium Modular Neck;
* Subject is willing and able to complete required study visits or assessments through the 10 year postoperative follow-up schedule;
* Subject is implanted with WMT or MPO head, cup and liner.

Newly or previously implanted bilateral subjects can have both Total Hip Arthroscopy enrolled in the study provided: 1) the specified PROFEMUR® Preserve Femoral Stems and cobalt-chromium Modular Necks were implanted in both, 2) all other aspects of the Inclusion/Exclusion Criteria are satisfied, 3) enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and 4) the subject agrees to a second Informed Consent document specific to the second Total Hip Arthroscopy.

Previously implanted subjects who had undergone revision of any Total Hip Arthroscopy component including the PROFEMUR® Preserve Femoral Stem(s) or, cobalt-chromium Modular Neck will also be eligible to be considered for this study.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Subjects implanted with non-MicroPort or Wright Medical Technology components (femoral heads, acetabular shells, acetabular liners);
* Subjects implanted with a PROFEMUR® Preserve stem assembled to a Titanium Modular Neck;
* Subjects skeletally immature (less than 21 years of age) at time of primary Total Hip Arthroscopy surgery;
* Subjects have or had an overt infection at the time of implantation;
* Subjects have or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation;
* Subjects have or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at time of implantation;
* Subjects have or had inadequate neuromuscular status (e.g., prior paralysis, fusion and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable;
* Subject has neuropathic joints;
* Subject has hepatitis or HIV infection;
* Subject has a neurological or musculoskeletal disease that may adversely affect gait or weight-bearing;
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol;
* Subjects unwilling or unable to sign the Informed Consent document;
* Subjects with documented substance abuse issues;
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study;
* Subjects who are incarcerated or have pending incarceration.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-arm, single-center, prospective follow-up study with consecutively enrolled newly or previously implanted subjects with the PROFEMUR® Preserve Femoral Stem(s) and CoCr (cobalt-chromium) Modular Neck combined with other Wright Medical Technologies (WMT) or MPO (MicroPort) THA (Total Hip Arthroscopy) components including acetabular shells, acetabular liners and femoral heads.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to evaluate component survivorship of the PROFEMUR® Preserve Femoral Stem and CoCr Modular Neck out to 10 years follow-up. | 10 years
  Percentage of hips survived with no revision or replacement at 10-year.

SECONDARY OUTCOMES:
To determine the cumulative incidence of component revision of the PROFEMUR® Preserve Femoral Stem and CoCr Modular Neck at specified intervals out to 10 years follow-up. | Time Frame: 2-5 years, 5-7 years, and 10 years
  Percentage of hips that were revised or replaced at each of the intervals namely for Early (2-5 years), midterm (5-7 Year), and long-term (10-year) evaluation.
To characterize functional scores, as assessed by Oxford Hip and EQ-5D-3L scores. | Time Frame: 2-5 years, 5-7 years, and 10 years
  The study will be reporting the final Oxford Hip score, which is a summary over 12 items. Each of these items is 5-level Likert scale such as from 'not at all' to 'totally'. EQ-5D-3L data will be summarized over 5 domains, namely, mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 3 levels: no problems, some problems, and extreme problems.
To evaluate the presence and the zones of radiolucencies surrounding the implanted femoral components. | 2-5 years, 5-7 years, and 10 years
  Radiolucencies are described around 7 zones and we will be reporting the number of hips with radiolucencies present at a given zone.
To characterize of adverse events and adverse device effects. | 2-5 years, 5-7 years, and 10 years
  Adverse Events will be summarized as the total number of Adverse Events (AE), Adverse Device Effect (ADE) by grade, severity, and relationship to the device and surgery. Number of patients experiencing such AEs and ADEs will be also provided.

CONTACTS AND LOCATIONS:
Overall Officials: Manel Ribas, MD, Principal Investigator — Hospital Universitari Dexeus
Locations (1):
- Dr. Manel Ribas, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No